CLINICAL TRIAL: NCT03771040
Title: A Prospective, Multicenter, Randomised, Double-blind, Placebo-controlled, Phase 3 Study to Compare the Efficacy and the Safety of Masitinib Versus Placebo in the Treatment of Patients With Severe Uncontrolled Asthma and Elevated Eosinophil Levels
Brief Title: Masitinib in the Treatment of Patients With Severe Uncontrolled Asthma and Elevated Eosinophil Levels
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AB14001
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-04

CONDITIONS: Asthma
Keywords: Severe persistent asthma; Eosinophil; Tyrosine kinase inhibitor
MeSH Terms: conditions — Asthma | interventions — masitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Masitinib (titration to 6.0 mg/kg/day) (Experimental): Participants receive masitinib (3.0 mg/kg/day), given orally twice daily, with a dose escalation to 4.5 mg/kg/day after 4 weeks of treatment, followed by dose escalation to 6.0 mg/kg/day after 4 weeks of treatment. Each ascending dose titration is subjected to a safety control.
  Interventions: Drug: Masitinib
- Placebo (Placebo Comparator): Participants receive matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Masitinib
  Other Names: AB1010
  Arms: Masitinib (titration to 6.0 mg/kg/day)
Drug: Placebo
  Other Names: Placebo Oral Tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of masitinib (6 mg/kg/day) in severe persistent asthma, uncontrolled with high dose of inhaled corticosteroid and with elevated eosinophil levels.

DETAILED DESCRIPTION:
Masitinib is a selective tyrosine kinase inhibitor. It is known that activation of inflammatory cells, such as mast cells, and fibrous tissue remodeling are associated with c-Kit, Lyn and PDGFR kinase signaling pathways; all key targets of masitinib. This is a multicenter, double-blind, randomized, parallel-group (ascending dose titration of masitinib to 6.0 mg/kg/day and matching placebo), comparative study of oral masitinib in the treatment of patients with severe asthma, uncontrolled with high dose of inhaled corticosteroid and with elevated eosinophil levels. Eligible patients will be treated during at least 48 weeks.

ELIGIBILITY:
Main inclusion criteria include:

* Patients with a physician diagnosis of persistent asthma for at least 12 months based on Global Initiative for Asthma (GINA) 2009 Guidelines whose asthma is partially controlled or uncontrolled on inhaled corticosteroids (ICS) / long-acting beta2-agonists (LABA) combination therapy.
* Patient with elevated eosinophil level related to asthma at baseline: ≥0.15 K/uL or patient with eosinophil level ≥0.15 K/uL related to asthma demonstrated in the year prior to screening
* Non-smoker patient for at least one year and with a prior tobacco consumption <10 packs/year

Main exclusion criteria include:

* Female patient who is pregnant or lactating
* Asthmatic patient still exposed to allergens or to triggering factors influencing asthma control
* Chronic obstructive pulmonary disease and/or other lung diseases impairing Pulmonary Function Tests
* Within 12 weeks prior to screening, patient who received oral corticosteroids for any other reason than to treat severe asthma exacerbation (patients needing long term corticosteroids intake to control basal asthma condition)
* Patient with history of acute infectious sinusitis or respiratory tract infection within 4 weeks prior to screening visit
* Patient with active lung disease other than asthma (e.g. chronic bronchitis)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Severe asthma exacerbation rate | Duration of patient treatment exposure, assessed until withdrawal from study, study completion date, or for a maximum of 60 months
  The number of severe asthma exacerbations over time frame of outcome measure

SECONDARY OUTCOMES:
Asthma exacerbation rate | Duration of patient treatment exposure, assessed until withdrawal from study, study completion date, or for a maximum of 60 months
  The number of asthma exacerbations over time frame of outcome measure
Asthma Control Questionnaire (ACQ) | 48 weeks
  Asthma Control Questionnaire (ACQ)
  * Type of questionnaire-description: A simple questionnaire to measure the adequacy of asthma control and change in asthma control which occurs either spontaneously or as a result of treatment.
  * Number of items: 7 items; 1 week recall (for items on symptoms and rescue inhaler use)
  * Number of domains & categories: ACQ has a multidimensional construct assessing symptoms (5 items--self-administred) and rescue inbronchodilator use (1 item-self-administered), and FEV1% (1 item) completed by clinic staff
  * Scaling of items: 7-point scale (0=no impairment, 6= maximum impairment for symptoms and rescue use; and 7 categories for FEV1%). Scores range between 0 (totally controlled) and 6 (severely uncontrolled).

CONTACTS AND LOCATIONS:
Overall Officials: Lavinia Davidescu, MD, PhD, Principal Investigator — University of Medicine and Pharmacy Oradea, Oradea, Romania.
Locations (5):
- Centro Respiratorio Quilmes, Buenos Aires, Argentina
- Sarawak General Hospital, Kuching, Malaysia
- Clínica Universidad de los Andes, Miraflores, Peru
- The Philippine Heart Center, Quezon City, Philippines
- National institute of phthisiology and pulmonology named after F.G. Yanovsky NAMS of Ukraine, Kiev, Ukraine

IPD SHARING:
Plan to Share IPD: No